CLINICAL TRIAL: NCT03992092
Title: Comparison of Video Stylet to Flexible Bronchoscopy for Intubation of Patients With Potential Cervical Spine Injury
Brief Title: Video Stylet vs. Flexible Bronchoscopy for C-Spine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Timothy Turkstra, Associate Professor and Staff Anesthesiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ReDa 7685
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Intubation;Difficult; Intubation Complication
Keywords: cervical spine injury

STUDY DESIGN:
Intervention Model Description: Parallel randomised controlled trial
Who Masked: Participant, Care Provider
Masking Description: Participants will be blinded, as will Anesthesiologist providing care, but the investigator who performs the intubation will be aware of the intubation technique he used. Similarly, the Radiologist measuring the C-spine movement will be able to see the device on the fluoroscopic images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C-Mac VS (Experimental): Intubation using the C-MAC Video Stylet
  Interventions: Device: C-MAC VS
- FB (Active Comparator): Intubation using the Flexible Bronchoscope
  Interventions: Device: Flexible Bronchoscopy

INTERVENTIONS:
Device: C-MAC VS — C-MAC Video Stylet
  Arms: C-Mac VS
Device: Flexible Bronchoscopy — Flexible Bronchoscopy
  Arms: FB

SUMMARY:
Comparison of cervical spine movement during intubation with the C-MAC Video Stylet to Flexible Bronchoscopy

DETAILED DESCRIPTION:
Elective surgical patients who require intubation will be randomised to one of 2 groups:

1. C-MAC Video Stylet
2. Flexible Bronchoscopy During intubation, fluoroscopy will be recorded for later analysis to determine the amount of cervical spine movement during the intubation process.

The intubation will also be timed to determine the duration of the intubation process.

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgery requiring oral intubation
* undergoing elective non-cardiac surgery
* American Society of Anesthesiologists physical status 1-3
* age 18-80 years

Exclusion Criteria:

* gastro-esophageal reflux disease
* body mass index > 35 kg/m2
* possibility of pregnancy
* previous neck surgery
* unstable C-spine
* known or predicted difficult airway.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to Intubation | Concurrent, during the intubation
  Duration of Intubation

SECONDARY OUTCOMES:
C-Spine Movement | Concurrent, during the intubation
  Degrees of C-Spine Movement as measured via Fluoroscope
Sore Throat | 24-48 hours post-op.
  Sore Throat rated as none, mild, moderate, or Severe
Vocal Changes | 24-48 hours post-op.
  Vocal Changes rated as none, mild, moderate, or Severe
Ease of Intubation | Concurrent, during the intubation
  Duration of Intubation, scored on a 100 mm VAS

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Turkstra, MD, Principal Investigator — LHSC
Locations (1):
- University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No